CLINICAL TRIAL: NCT04560101
Title: Motor and Non-motor Symptoms in Patients With Cervical Dystonia and the Effect of Treatment With Botulinum Toxin A
Brief Title: Motor and Non-motor Symptoms in Cervical Dystonia
Acronym: Royal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Giovanni Fabbrini, Full Professor of Neurology, University of Roma La Sapienza
Other Study IDs: 5491
Record Dates: First submitted 2020-09-09; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Dystonia, Focal
Keywords: depression; anxiety; sleep; cognitive
MeSH Terms: conditions — Dystonic Disorders; Depression; Anxiety Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: botulinum toxin A — Intramuscolar injection of botulinum toxin in affected muscles

SUMMARY:
In this monocenter, observational, non-interventional, prospective, open label study investigators will enrol 43 CD patients from the outpatient Movement Disorders Clinic of the Department of Human Neurosciences, Sapienza University of Rome.

As this is a non-interventional study, no diagnostic, therapeutic or experimental intervention is involved. Subjects will receive clinical assessments, medications and treatments solely as determined by their study physician. The BoNT-A injection will be performed in CD patients at baseline.

As this is an observational, non-interventional study, the injection protocol for BoNT-A treatment is upon physicians' decision. All CD patients will undergo up to three evaluations of motor and non-motor symptoms: before (baseline) and 1 month and 3 months after botulinum toxin treatment. Both evaluations will be carried out under the same conditions. Motor symptoms will be assessed in all CD using the Comprehensive Cervical Dystonia Rating scale (CCDRS) (Comella et al, 2015). Non-motor symptoms including psychiatric, psychological and sleep disorders will be investigated. Psychiatric symptoms will be assessed with CCDS, Hamilton Rating Scale for Anxiety (HAM-A) and the Hamilton Rating Scale for Depression (HAM-D); the psychological symptoms will be assessed with the demoralization scale (Kissane et al, 2004) and the Italian Perceived Disability Scale (Innamorati et al,2009). Sleep disorders will be investigated with the Pittisburg Sleep Quality Index (PSQI) (Buysse et al, 1989).

DETAILED DESCRIPTION:
Cervical dystonia (CD) is a focal dystonia, characterized by sustained muscle contractions of the neck causing repetitive movements, or abnormal postures. The muscles' activation pattern may lead to neck rotation (torticollis), flexion (anterocollis), extension (retrocollis), or head tilt (laterocollis) or a combination of these. Patients with CD may also have head tremor.

In addition to motor symptoms, CD patients may have non-motor features including psychiatric disturbances, sleep difficulties, cognitive impairment and neck pain.

The first line of treatment for CD is botulinum toxin-A (BoNT-A) injection therapy administered approximately at every 12 weeks. Several studies showed that one month after BoNT-A treatment there is an improvement of motor symptoms in the majority of CD patients. Conversely, regarding the effect of BoNT-A on non-motor symptoms previous studies in CD focused only on the possible effect on depressive symptoms and on neck pain.

No study has so far investigated whether the treatment with BoNT-A may improve non-motor symptoms in CD, including psychological aspects, such as demoralization and perceived disability.

Main aim of this study is therefore to assess the effect of botulinum neurotoxin type A (BoNT-A) treatment on motor and non-motor symptoms, including psychiatric and psychological symptoms (anxiety, depression, demoralization, perceived disability) and sleep. To this aim CD patients will be re-tested at 1 month and at 3 months after the treatment with BoNT-A. Investigators will also assess a possible relationship between the improvements of motor symptoms with that of non-motor symptoms at 1 month and at 3 months after BoNT-A treatment and the frequency and severity of non-motor symptoms in a large population of CD patients.

To see whether non-motor symptoms in CD are the consequence of motor symptoms, investigators will compare the severity of non-motor symptoms with the severity of motor symptoms, as well as with the different clinical patterns of CD and with the presence or absence of head tremor.

ELIGIBILITY:
Inclusion Criteria:

* Cervical dystonia patients (primary dystonia).
* BoNT-A naïve or pre-treated with any BoNT-A product.
* Signed informed consent prior to participation in the study. If previously treated with any BoNT-A, at least a 3-4 months interval between last injection and inclusion.

Exclusion Criteria:

* - All secondary causes of dystonia (e.g. parkinsonian syndromes, or exposition of dopamine receptor blocking drugs) will be excluded.
* Major psychiatric disorders.
* Sensitivity to BoNT-A or to its excipients
* Other contraindications as given in the local SmPC for BoNT-A
* Pregnant & lactating women

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of Cervical dystonia
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes in depression scores from baseline to month 1 and 3 | From baseline to month 1 and 3 after treatment
  Changes in the Hamilton Rating Scale for depression (HAM-D) before and after three months from treatment
Changes in anxiety scores from baseline to month 1 and 3 | From baseline to month 1 and 3 after treatment
  Changes in the Hamilton Rating Scale for anxiety (HAM-A) before and after three months from treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Fabbrini, MD, Principal Investigator — Depatment Human Neurosciences Sapienza University of Rome
Locations (1):
- Department of Human Neurosciences, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
Single center study

REFERENCES:
- [Result] Fabbrini G, Berardelli I, Moretti G, Pasquini M, Colosimo C, Berardelli A. Nonmotor symptoms in adult-onset focal dystonia: psychiatric abnormalities. Mov Disord. 2011 Aug 1;26(9):1765-6. doi: 10.1002/mds.23668. Epub 2011 Mar 25. No abstract available. PMID 21442656
- [Result] Berardelli I, Ferrazzano G, Pasquini M, Biondi M, Berardelli A, Fabbrini G. Clinical course of psychiatric disorders in patients with cervical dystonia. Psychiatry Res. 2015 Sep 30;229(1-2):583-5. doi: 10.1016/j.psychres.2015.07.076. Epub 2015 Jul 29. PMID 26239770
- [Result] Conte A, Berardelli I, Ferrazzano G, Pasquini M, Berardelli A, Fabbrini G. Non-motor symptoms in patients with adult-onset focal dystonia: Sensory and psychiatric disturbances. Parkinsonism Relat Disord. 2016 Jan;22 Suppl 1:S111-4. doi: 10.1016/j.parkreldis.2015.09.001. Epub 2015 Sep 3. PMID 26360238
- [Result] Ferrazzano G, Berardelli I, Conte A, Suppa A, Fabbrini G, Berardelli A. Interoceptive sensitivity in patients with cervical dystonia. Parkinsonism Relat Disord. 2017 Nov;44:129-132. doi: 10.1016/j.parkreldis.2017.08.019. Epub 2017 Aug 16. PMID 28827008
- [Result] Ferrazzano G, Berardelli I, Conte A, Baione V, Concolato C, Belvisi D, Fabbrini G, Defazio G, Berardelli A. Motor and non-motor symptoms in blepharospasm: clinical and pathophysiological implications. J Neurol. 2019 Nov;266(11):2780-2785. doi: 10.1007/s00415-019-09484-w. Epub 2019 Jul 29. PMID 31359200
- [Result] Berardelli I, Ferrazzano G, Belvisi D, Pompili M, Fabbrini G. Psychiatric disorders in blepharospasm: A 10-year follow-up study. Psychiatry Res. 2020 Aug;290:113092. doi: 10.1016/j.psychres.2020.113092. Epub 2020 May 26. No abstract available. PMID 32505028
- [Result] Ferrazzano G, Berardelli I, Belvisi D, De Bartolo MI, Di Vita A, Conte A, Fabbrini G. Awareness of Dystonic Posture in Patients With Cervical Dystonia. Front Psychol. 2020 Jun 23;11:1434. doi: 10.3389/fpsyg.2020.01434. eCollection 2020. PMID 32655462
- [Result] Berardelli I, Ferrazzano G, Belvisi D, Baione V, Fabbrini G, Innamorati M, Berardelli A, Pompili M. Suicidal ideation, hopelessness, and affective temperament in patients with blepharospasm. Int J Psychiatry Clin Pract. 2021 Nov;25(4):344-349. doi: 10.1080/13651501.2020.1790613. Epub 2020 Jul 15. PMID 32669012